CLINICAL TRIAL: NCT06666595
Title: Clinical Outcome of Subcrestal Short Implant Versus Crestal Standard Length Implant to Retain Kennedy Class 1 Removable Partial Denture: A Split-mouth Study
Brief Title: Short Implant Versus Crestal Standard Length Implant to Retain Class 1 Removable Partial Denture.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Collaborators: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed El-Sawy, lecturer, Department of Prosthetic Dental Sciense, principle investigator, Menoufia University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: ADMNF-00701124
Record Dates: First submitted 2024-10-26; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Bone Loss; Partial Edentulism Class 1
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subcrestal short implant (Active Comparator): Evaluation the amount of bone loss after one, two, and three years of function.
  Interventions: Procedure: Titanium dental implant (Conical SPI, Vitronix, Italy), Medical device that interfaces with the jawbone to support a dental prosthesis.
- crestal standard length implant (Active Comparator): Evaluation the amount of bone loss after one, two, and three years of function.
  Interventions: Procedure: Titanium dental implant (Conical SPI, Vitronix, Italy), Medical device that interfaces with the jawbone to support a dental prosthesis.

INTERVENTIONS:
Procedure: Titanium dental implant (Conical SPI, Vitronix, Italy), Medical device that interfaces with the jawbone to support a dental prosthesis. — Placement of titanium dental implant to retain and support Kennedy class 1 removable partial denture (RPD).The implant fuses with the bone through a process called osseointegration.

SUMMARY:
Objective: To report the implant survival rates, clinical, and radiographic outcomes of subcrestal short implant versus crestal standard length implant supported removable partial denture (RPD).

DETAILED DESCRIPTION:
30 individuals with at least 2 adjacent missing teeth bilaterally were included.to support class Ι RPD with conventional loading protocol were chosen for this research. Each participant received 2 implants in a split mouth design, one side received 1 subcrestal short implant and the contralateral side crestal standard length implant. Plaque index (PI), bleeding on probing (BOP), probing depth (PD), radiographic crestal bone level (CBL) and implant survival rate were evaluated. at implant placement (T0), restoration delivery (T1), and 3-year follow-up after loading (T2). MBL was calculated as the change in distance from the implant-abutment interface to the first radiographically visible bone-implant contact. A repeated-measures mixed ANOVA followed by a paired Student's t-test with the Bonferroni correction was used for statistical analysis. p < 0.05 was considered statistically significant

ELIGIBILITY:
Inclusion Criteria

* adult patients aged 50 years or older with class 1 RPD with missing mandibular molars at least and complaining from instability of the prosthesis were recruited.
* Medical history revealed no contraindication to implant therapy.
* Patients have an amount of bone nearly equal to 8 mm length above the inferior alveolar canal to receive a 6 mm short implant with 2 mm subcrestal to the bone level with sufficient bone width ≥ 8mm on one side and an amount of bone equal to or more than 8 mm to receive a standard-length implant of 7.5, 9, or 10.5 mm placed at crestal bone level with sufficient bone width ≥ 8mm on the contralateral side which was examined by CBCT.

Exclusion Criteria:

* Presence of active infection or inflammation in the areas intended for implant placement; *systemic diseases such as diabetes.
* Pregnant and lactating patients.
* Habit of severe bruxism or clenching.
* Treatment with therapeutic radiation to the head within the past 12 months.
* Treatment with bisphosphonate within the past 12 months.
* More than 10 cigarettes/day smoking habit.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2025-04-20 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Bone loss | 3 years
  Evaluation of crestal bone loss around implants will be performed by periapical digital radiograph using parallel technique to avoid distortion or elongation to the image.

SECONDARY OUTCOMES:
Plaque index (PI) | 3 years
  Evaluation of PI around implants were assessed by using a numerical recording of BI (present = 1; absent = 0), PI (present = 1; absent = 0), as well as PD. With the use of a plastic periodontal probe (Hu-Friedy, Chicago, Illinois).
Bleeding on probing (BOP) | 3 years
  Evaluation of BOP around implants were assessed by using a numerical recording of BOP (present = 1; absent = 0), PI (present = 1; absent = 0), as well as PD. With the use of a plastic periodontal probe (Hu-Friedy, Chicago, Illinois).

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammed A. El-Sawy, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No
Up on reasonable request from the corresponding author